CLINICAL TRIAL: NCT07282444
Title: Collaborative Oncology Between Radiologists and Radiation Oncologists for the Evaluation of Contoured Targets (CORRECT)
Brief Title: A New Way to Share Radiation Therapy Plans Between Doctors, CORRECT Trial
Acronym: CORRECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00141160; U34CA297499 (NIH); UG1CA189824 (NIH); P30CA012197 (NIH); NCI - 2025-07036 (Other: NCI Trial Identifier); WF-2402CD (Other: Lead Organization Identifier); WF-2402CD (Other: DCP Identifier); WF-2402CD (Other: CTEP Identifier)
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lung Carcinoma; Head and Neck Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Educational Status; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: No Data Available
Masking Description: No Data Available
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (CORRECT workflow) (Experimental): ROs and radiologists receive training on the use of the CORRECT workflow and practice with test cases. ROs and radiologists then use the CORRECT workflow with patient cases for 12 months.
  Interventions: Behavioral: Training and Education; Other: Communication Intervention; Other: Survey Administration; Other: Interview; Other: Electronic Health Record Review

INTERVENTIONS:
Behavioral: Training and Education — Receive training and practice cases on CORRECT workflow
Other: Communication Intervention — Use CORRECT workflow
Other: Survey Administration — Ancillary studies
Other: Interview — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial tests a new way to share radiation therapy plans using the Collaborative Oncology between Radiologists and Radiation oncologists for the Evaluation of Contoured Targets (CORRECT) workflow to improve communication and collaboration between radiation oncologists (ROs) and radiologists when determining cancer targets for radiation treatment. Systemic barriers limit critical communication between radiation oncologists and radiologists and can lead to both under and overdosing of radiation therapy (RT) tumor targets and failures to properly interpret post-treatment imaging. The limited formal diagnostic radiology training of many providers can make differentiating normal from disease imaging findings during target determination difficult, especially in complex disease sites like the lung, head, and neck. Inaccurate target determination may result in cancer return, excess toxicity, or both. Likewise, radiologists who cannot access prior RT plans may mistake expected RT changes for recurrent cancer or overlook true progression. The CORRECT workflow was developed by ROs and radiologists to address RO-radiology communication barriers by facilitating sharing of comprehensive RT target contours during RT planning. The CORRECT workflow begins with the normal process of RO target contouring. Computed tomography (CT) images are then fused with RT targets and pushed to a pre-designated Picture Archiving and Communications System (PACS) software folder accessible by the radiology department. The radiologist can then review the fused images at their chosen time and annotate images to indicate potential deviations (e.g., not avoiding normal tissue or not including all tumor). The RO reviews the annotated images and decides if any changes to treatment targets are needed for the final treatment plan. Through this independent, asynchronous review of high-quality images, CORRECT overcomes many of the limitations of existing communication methods between RO-radiologist, fostering a more collaborative, efficient, and precise approach to cancer treatment planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the feasibility of the CORRECT workflow, defined as the return of radiology feedback via CORRECT within 2 business days from receipt of initial RT targets.

SECONDARY OBJECTIVES:

I. To further assess the feasibility of the CORRECT workflow as measured by 1) time (in business days) required to install the information technology (IT) application at each practice, 2) the number and proportion of cases per practice with reports of technical issues requiring centralized IT or CORRECT study team assistance, 3) percentage of approached patients who declined consent.

II. To assess ROs and radiologists' perceptions of acceptability, appropriateness and feasibility of the CORRECT workflow using the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM), along with the acceptability of CORRECT workflow training.

III. To identify facilitators and barriers to radiation oncology-radiology standard of care collaboration, CORRECT workflow implementation, and participation in the future trial using a qualitative interview.

OUTLINE:

ROs and radiologists receive training on the use of the CORRECT workflow and practice with test cases. ROs and radiologists then use the CORRECT workflow with patient cases for 12 months

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE: Must provide radiation therapy for ≥ 3 patients per month with lung cancer or head & neck cancer
* PRACTICE: At least one radiation oncologist and one radiologist (in house, contracted, etc.) at the practice willing to participate, but may have multiple participants at the practice
* PRACTICE: Radiation oncologist/radiologist team must use Picture Archiving and Communication System (PACS) software at this practice
* RADIATION ONCOLOGIST (NON-PATIENT): Must have been in independent practice (i.e., performing duties without preceptor oversight) for a minimum of six months
* RADIATION ONCOLOGIST (NON-PATIENT): Must treat lung and/or head & neck cancer patients with curative intent radiation therapy
* RADIATION ONCOLOGIST (NON-PATIENT): Willing and able to participate in 15 minutes of mandatory virtual CORRECT training
* RADIATION ONCOLOGIST (NON-PATIENT): Willing to participate in a 30-minute interview, if selected at the end of the study
* RADIOLOGIST (NON-PATIENT): Must have been in independent practice (i.e., performing duties without preceptor oversight) for a minimum of six months
* RADIOLOGIST (NON-PATIENT): Agree to review pre-treatment radiation therapy targets during the course of the study duration (approximately 12 months). Willing and able to participate in 15 minutes of mandatory virtual CORRECT training
* RADIOLOGIST (NON-PATIENT): Willing to participate in a 30-minute interview, if selected at the end of the study
* PATIENT: Must have any stage of clinically diagnosed lung or head & neck (HN) cancer
* PATIENT: Planned treatment with curative intent definitive RT (with or without other treatments). Curative intent RT must be documented in the electronic medical record (EMR) by the treating radiation oncologist
* PATIENT: Must be expected to be treated by a radiation oncologist participating in this study
* PATIENT: Must be 18 years or older

Exclusion Criteria:

* PRACTICE: Participation by the Community Site or Minority/Underserved Community Site in another National Cancer Institute (NCI) Community Oncology Research Program (NCORP) Cancer Care Delivery Research (CCDR) U34-supported protocol funded in NCI fiscal year 2025 or later. (Note: WF- 2301CD CONNECT is exempt from this policy, as it was funded prior to NCI fiscal year 2025.)
* RADIATION ONCOLOGIST (NON-PATIENT): Planning to leave their position at this practice within the next 12 months
* RADIATION ONCOLOGIST (NON-PATIENT): Providing service on a temporary basis (i.e., locum tenens providers)
* RADIOLOGIST (NON-PATIENT): Planning to leave their position at this practice within the next 12 months
* RADIOLOGIST (NON-PATIENT): Providing service on a temporary basis (i.e., locum tenens providers)
* PATIENT: Unable to understand English or Spanish
* PATIENT: Early glottic larynx cancer planned for definitive RT alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
The return of radiology feedback via Collaborative Oncology between Radiologists and Radiation oncologists for the Evaluation of Contoured Targets (CORRECT) (feasibility) | Within 2 business days from receipt of initial radiation therapy (RT) targets
  If > 50% of patients have target feedback returned to the radiation oncologist within 2 business days, this workflow will be considered feasible in community practice.

SECONDARY OUTCOMES:
Time (in business days) required to install the information technology (IT) application | During study start-up prior to the enrollment of first patient case; up to 60 days after CIRB approval at the practice.
  Will be assessed at each practice as tracked on the CORRECT IT data form
The number and proportion of cases per practice with reports of technical issues requiring centralized IT or CORRECT study team assistance | During RT planning for each patient; over the 9 months of of patient accrual
  Will be assessed at each practice as tracked on the CORRECT IT data form.
Percentage of approached patients who declined consent | During screening and enrollment over the 9 months of patient accrual
  Will be assessed at each practice as tracked on the Patient Refusal form.
Acceptability of the CORRECT workflow. | Up to 2 months after patient enrollment has concluded
  Will be assessed using the Acceptability of Intervention Measure. Will be collected on the post-study radiation oncologist/radiologist survey. Scale has four items measured on a Likert scale from 1 (completely disagree) to 5 (completely agree). The four items are averaged to obtain a final score.
Appropriateness of the CORRECT workflow | Up to 2 months after patient enrollment has concluded
  Will be assessed using the Intervention Appropriateness Measure. Will be collected on the post-study radiation oncologist/radiologist survey. Scale has four items measured on a Likert scale from 1 (completely disagree) to 5 (completely agree). The four items are averaged to obtain a final score.
Feasibility of the CORRECT workflow | Up to 2 months after patient enrollment has concluded
  Will be assessed using the Feasibility of Intervention Measure. Will be collected on the post-study radiation oncologist/radiologist survey. Scale has four items measured on a Likert scale from 1 (completely disagree) to 5 (completely agree). The four items are averaged to obtain a final score.
Facilitators and barriers to radiation oncology-radiology standard of care collaboration, CORRECT workflow implementation, and participation in the future trial | Up to 2 months after patient enrollment has concluded
  Will be identified using qualitative interviews using the radiation oncologist/radiologist interview guide.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, Study Chair — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wfusm.edu
URL: http://nctn-data-archive.nci.nih.gov/